CLINICAL TRIAL: NCT03979443
Title: Finnish Trial on Practices of Anterior Cervical Decompression and Fusion (FACADE): A Protocol for a Prospective Randomized Non-inferiority Trial Comparing Outpatient vs. Inpatient Care
Brief Title: Finnish Trial on Practices of Anterior Cervical Decompression (FACADE) Comparing Outpatient vs. Inpatient Care
Acronym: FACADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Turku University Hospital (Other Government); Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Kimmo Lonnrot, Principal Investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1540/2019
Record Dates: First submitted 2019-06-04; First posted 2019-06-07 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Cervical Radiculopathy
Keywords: Anterior cervical decompression and fusion; cervical fusion; cervical spine; spinal surgery; outpatient care; randomized controlled trial; Protocol
MeSH Terms: conditions — Radiculopathy; Klippel-Feil Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatient (No Intervention): patients staying in the hospital for 1-3 nights after surgery
- Outpatient (Active Comparator): discharge on the day of the surgery, usually within 6-8 hours after procedure
  Interventions: Procedure: Discharge on the day of surgery

INTERVENTIONS:
Procedure: Discharge on the day of surgery — Patient discharge on the day of the surgery, usually within 6-8 hours after procedure
  Arms: Outpatient

SUMMARY:
FACADE is a prospective, randomized, controlled, parallel group non-inferiority trial comparing the traditional hospital surveillance (inpatient, patients staying in the hospital for 1-3 nights after surgery) to outpatient care (discharge on the day of the surgery, usually within 6-8 hours after procedure) in patients who have undergone anterior cervical decompression and fusion (ACDF) procedure.

DETAILED DESCRIPTION:
To determine whether early discharge (outpatient care) is noninferior to inpatient care, the investigators will randomize 104 patients to these two groups and follow them for 6 months using the Neck Disability Index (NDI) as the primary outcome. The investigators expect that early discharge is not significantly worse (inferior) than the current care in terms of change in NDI. Noninferiority will be declared if the mean improvement for outpatient care is no worse than the mean improvement for inpatient care, within statistical variability, by a margin of 17.3%. The investigators hypothesize that a shorter hospital stay results in more rapid return to normal daily activities, shorter duration of sick leave and decreased secondary costs to health care system. Secondary outcomes in the study are arm pain and neck pain using the Numeric Rating Scale, operative success (Odom's criteria), patient's satisfaction to treatment, general quality of life (EQ-5D-5L), work ability score (WAS), sickness absence days, return to previous leisure activities, and complications.

Patients who are eligible for the trial, but are not willing to undergo randomization, will be asked to be included in a simultaneous, pragmatic follow-up cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Cervical radiculopathy syndrome (CRS) unresponsive to non-operative treatment for at least six weeks or with severe progressive signs and symptoms of nerve root compression during conservative treatment of shorter duration.
2. CRS is defined as pain, paresis or paresthesia in corresponding nerve root distribution areas of C5, C6, C7 or C8.
3. Nerve root stenosis determined by magnetic resonance imaging at treatment level correlating to CRS/symptoms
4. Neck Disability Index score ≥30 out of 100
5. Age between 18 to 62 years
6. No previous cervical operations
7. Currently employed
8. No co-morbidities causing a need for a sick leave
9. Provision of informed consent from the participant
10. No contraindication for randomization in postoperative check (see below)

Exclusion Criteria:

1. MRI finding inconsistent with patient's symptoms
2. Diagnosed osteoporosis or permanent use of oral corticosteroids
3. ACDF operation requiring plate or cage fixation with screws
4. Active malignancy
5. American Society of Anesthesiologists Physical Status Classification system (ASA) 4 and 5 patients (seriously ill patients)
6. Pregnancy
7. Abundant use of alcohol, drugs or narcotics
8. No possibility to be accompanied by an adult person over the first postoperative night after the surgery
9. Insufficient Finnish language skills
10. Distance to the closest hospital emergency more than 60 min

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Neck Disability Index at 6 months after operation | Before and up to 6 months after operation
  Neck disability Index scale score ranges from 0 to 100%. Score 0 indicates no disability as score 100% indicates worst possible disability.

SECONDARY OUTCOMES:
Change from baseline Numeric rating scale on arm pain at six months after operation | Before and up to 6 months after operation
  Numeric rating scale ranges from 0 to 10, where 0 indicates no pain and 10 indicates worst possible pain
Change from baseline Numeric rating scale on neck pain at six months after operation | Before and up to 6 months after operation
  Numeric rating scale ranges from 0 to 10, where 0 indicates no pain and 10 indicates worst possible pain
Rate of returning to previous leisure activities after operation | Before and up to 6 months after operation
  Before the operation, participants will be asked to name the most important daily leisure activity they are not able to perform because of the disease. At each follow-up time point (Table 2), participants will be asked to respond to the following question: "Have you been able to return to your leisure activity?" ("yes" or "no")
Change from baseline Work Ability Score (WAS) at six months after operation | Before and up to 6 months after operation
  Numeric rating score ranges from 0 to 10, where 0 indicates that participant is completely incapable to work and 10 indicates participants work ability at its best
The duration of sick leave | Before and after operation
  the number of sickness absence days from work both before and after the operation. The number of sickness absence days will be treated as a continuous variable

OTHER OUTCOMES:
Change from baseline Euroqol 5 dimensional questionnaire of generic quality of life measurement (EQ-5D-5L) at six months after operation | Before and at 6 months after operation
  EQ-5D-5L descriptive score ranges from 0 (no problems in health state) to 25 (maximal problem in health state). EQ-5D-5L Visual analogic score (VAS) ranges form 0 (the worst health) to 100 (the best health) assessed by participant.
Patient satisfaction to treatment | at six months after operation
  patients' global assessment of satisfaction to the treatment at six months after operation with this question: "If you were to choose again, would you choose an operative treatment?" ("yes" or "no").
Operative success | at one week, one month, three months and six months after operation
  patient subjectively rates the perception of operative success from poor to excellent by the modified Odom's criteria. the first and second categories ('excellent' and 'good') as a successful outcome of the operation and conversely, last two categories ('fair' and 'poor') as an unsuccessful outcome.
Rate of complications and adverse effects | From operation up to six months postoperatively
  The rate of complications related to intervention or operation in both group after operation

CONTACTS AND LOCATIONS:
Overall Officials: Kimmo Lonnrot, MD, PhD, Principal Investigator — Senior neurosurgeon at Helsinki Univ. Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) is available upon request when General Data Protection Regulation (GDPR) and guiding legislation regulations are fulfilled.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study protocol and Statistical Analysis Plan (SAP) will be published after the study has started. Other document will be available as study proceeds and after study is completed.
Access Criteria: Data access request will be reviewed by FACADE steering group. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Lonnrot K, Taimela S, Satopaa J, Saarenpaa I, Leinonen V, Kivelev J, Silvasti-Lundell M, Forster J, Pitkanen M, Raj R, Kauppinen M, Westermarck R, Jahromi BR, Koski-Palken A, Seppala M, Kivipelto L, Antinheimo J, Korja M, Czuba T, Jarvinen TLN. Ambulatory Care vs Overnight Hospitalization After Anterior Surgery for Cervical Radiculopathy: The FACADE Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2447459. doi: 10.1001/jamanetworkopen.2024.47459. PMID 39602120
- [Derived] Lonnrot K, Taimela S, Toivonen P, Aronen P, Koski-Palken A, Frantzen J, Leinonen V, Silvasti-Lundell M, Forster J, Jarvinen T; FACADE investigators. Finnish Trial on Practices of Anterior Cervical Decompression and Fusion (FACADE): a protocol for a prospective randomised non-inferiority trial comparing outpatient versus inpatient care. BMJ Open. 2019 Nov 26;9(11):e032575. doi: 10.1136/bmjopen-2019-032575. PMID 31772100

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT03979443/SAP_000.pdf